CLINICAL TRIAL: NCT07066150
Title: Efficacy of Marula Oil-Derived Ceramide Cream in Improving Skin Barrier Function: A Clinical Evaluation
Brief Title: A Clinical Evaluation of Marula-Derived Ceramide Cream on Skin Barrier Function Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chicmax Cosmetic Co., Ltd. (Industry)
Collaborators: SGS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: QDCPCH2500065-02-CN
Record Dates: First submitted 2025-06-19; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis (AD); Psoriasis; Acne Vulgaris; Contact Dermatitis; Photodamaged Skin; Ichthyosis; Xerosis Cutis
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis; Acne Vulgaris; Dermatitis, Contact; Ichthyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Marula Oil-Derived Ceramide NPs Cream Treatment Group (Experimental): The participants were requested to apply a cream containing 0.05% marula oil-derived ceramide NPs on their faces twice daily for 28 consecutive days.
  Interventions: Other: Apply a cream containing 0.05% marula oil-derived ceramide NPs

INTERVENTIONS:
Other: Apply a cream containing 0.05% marula oil-derived ceramide NPs — The participants were requested to apply a cream containing 0.05% marula oil-derived ceramide NPs on their faces twice daily for 28 consecutive days.

SUMMARY:
Previously, the investigators have demonstrated in vitro the excellent efficacy of marula oil-derived ceramide NPs in enhancing skin barrier function. The investigators's findings show that marula oil-derived ceramide NPs not only significantly reduces levels of inflammatory cytokines but also promotes the expression of key proteins in skin barrier integrity. These results suggest that marula oil-derived ceramide NPs may offer a more effective therapeutic option for skin barrier-disrupted diseases. Therefore, the investigators aim to further investigate the repair function of marula oil-derived ceramide NPs on the human epidermal barrier through a clinical trial.

DETAILED DESCRIPTION:
Marula oil, a botanical ingredient widely utilized in the cosmetics industry, has attracted significant attention due to its exceptional skin-beneficial attributes. Characterized by its richness in monounsaturated fatty acids, predominantly oleic acid, and antioxidants, marula oil exhibits potent moisturizing, anti-inflammatory, anti-aging, and antioxidant activities. Notably, despite sharing a similar fatty acid profile with olive oil, marula oil demonstrates tenfold greater resistance to lipid oxidation. Additionally, the fatty acid chain lengths of marula oil, spanning from C14 to C22, closely align with those of human skin ceramides, positioning it as an ideal precursor for the synthesis of plant-derived ceramide NPs.

Previously, the investigators has demonstrated in vitro that marula oil-derived ceramide NPs have excellent efficacy in enhancing skin barrier function. The investigators' findings show that marula oil-derived ceramide NPs not only significantly reduce levels of inflammatory cytokines but also promote the expression of key proteins in skin barrier integrity. These results suggest that marula oil-derived ceramide NPs may offer a more effective therapeutic option for skin barrier-disrupted diseases. Therefore, the investigators aim to further investigate the repair function of marula oil-derived ceramide NPs on the human epidermal barrier through a clinical trial.

Against this backdrop, the investigators aims to assess the efficacy of a marula oil-derived ceramide NPs cream in moisturizing, soothing, and repairing the skin barrier. A 28-day prospective study will be conducted on adult subjects, who will use the product as directed under standardized conditions. The investigation will also evaluate the suitability of the cream for sensitive skin, focusing on its non-irritating properties.

ELIGIBILITY:
Inclusion Criteria

* Healthy females aged 18 to 60 years
* Skin types: oily, combination oily, neutral, dry, or combination dry
* Ethnicity: Asian (Chinese)
* Sensitive skin confirmed by lactic acid stinging test screening
* Transepidermal water loss (TEWL) > 15 g/h/m² in one cheek area
* Stratum corneum moisture content <50 C.U. in one cheek area
* Visual redness score 3-6 per SGS standard atlas (0-9 scale, 0.5-point increment)
* Willingness to sign photo consent form
* No significant skin lesions, scars, or excessive facial/neck hair
* Ability to comply with protocol requirements and maintain consistent lifestyle

Exclusion Criteria Refusal to sign informed consent

* Unwillingness to comply with protocol requirements
* Concurrent participation in other clinical studies
* Cosmetic/drug use on assessment day
* Pregnancy or lactation (self-reported)
* Pharmacological treatment during study
* Infectious skin diseases or atopic dermatitis
* Skin abnormalities in assessment area (e.g., moles, telangiectasia)
* Skin peeling/cosmetic procedures within 3 months prior to enrollment
* Immunosuppressant therapy within 3 months prior to enrollment
* Systemic steroid treatment or phototherapy within 1 month prior to enrollment
* Use of topical medications/special efficacy cosmetics on target area within 2 weeks prior to enrollment
* Assessment area lesions interfering with measurements
* History of severe reactions to cosmetics, drugs, or light exposure
* Principal Investigator discretion of unsuitability

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of Transepidermal Water Loss (TEWL) Following Topical Facial Cream Application | Outcome assessments: baseline (Day 0), Day 7, and Day 28 (after 28 days of twice-daily cream application). Total study duration: 28 days.
  This study measures transepidermal water loss (TEWL) using a Tewameter (Tewameter® TM Hex) device. TEWL measurements are obtained from the standardized cheek area (left and right sides) at baseline (Day 0), 7 days after initiating twice-daily application of the topical facial cream (Day 7), and 28 days after initiation (Day 28). The primary outcome is the TEWL rate, quantified as grams per hour per square meter (g/h/m²).
Evaluation of Skin Hydration Following Application of a Topical Facial Cream | Outcome measures are assessed at baseline (Day 0), Day 7 (7 days after cream initiation), and Day 28 (28 days after cream initiation). Participants apply the cream twice daily throughout the 28-day study period.
  This clinical study evaluates stratum corneum hydration in adult participants using a Corneometer® CM 825 device. Standardized measurements of the designated cheek area (either left or right side, consistently applied for all participants) are performed to assess the primary parameter: stratum corneum moisture content, which is reported in Corneometer Units (C.U.). The study follows a structured protocol where the topical facial cream is applied twice daily as the investigational intervention, aiming to characterize its impact on skin hydration over the study period.
Evaluation of Erythema Severity Using a* Color Value in Facial Skin | Measurements at Baseline (Day 0), Day 7, and Day 28 during the 28-day intervention period.
  This clinical study quantifies facial erythema severity in adult participants by analyzing the CIELAB a* color value derived from VISIA CR 5.0 - captured images. The target assessment area is a standardized unilateral cheek region (consistently left or right as per pre - defined protocol). Measurements follow a structured protocol, with the primary outcome defined as the change in a* color value over time, which directly reflects erythema intensity modulation. All image acquisitions and a* value extractions adhere to validated VISIA CR 5.0 operating procedures to ensure data reliability.
Quantitative Assessment of Facial Erythema Area. | Outcome assessed at Baseline (Day 0), Day 7 , and Day 28 during 28-day study.
  This clinical study quantitatively assesses facial erythema area in adult participants using the VISIA CR 5.0 system's erythema analysis module. Erythema area percentage (%) is measured at a pre - defined standardized unilateral cheek region (consistently left or right, per protocol). Assessments follow the device's standard erythema detection mode under controlled, validated lighting conditions. The primary outcome is the change in erythema area percentage over the study period, with all measurements adhering to VISIA CR 5.0's validated operating procedures to ensure data reliability.
Effect of Topical Facial Cream on Skin Thickness. | Assessments at Baseline (Day 0), Day 7 , and Day 28 during 28-day intervention period.
  This clinical study evaluates the effect of a topical facial cream on skin thickness in adult participants. Using the Dermalab® Combo device, standardized measurements of epidermal and dermal thickness (μm) are performed at the zygomatic fat region of a pre - defined unilateral cheek (consistently left or right, per protocol). The primary outcomes are changes in epidermal thickness and dermal thickness over the study period, with all assessments following validated Dermalab® Combo operating procedures to ensure data reliability. The topical facial cream is applied as per the study protocol, and measurements adhere to a structured schedule to characterize its impact on skin thickness.
Effect of Topical Facial Cream on Skin Density | Outcome assessed at Baseline (Day 0), Day 7, and Day 28 during 28-day intervention period
  This clinical study evaluates the effect of a topical facial cream on facial skin density in adult participants. Using the Dermalab® Combo device, standardized measurements of skin density are performed at the zygomatic fat region of a pre-defined unilateral cheek (consistently left or right, per protocol). Skin density is quantified in device-specific arbitrary units, with all assessments following validated Dermalab® Combo operating procedures to ensure data reliability. The primary outcome is the change in skin density over the study period, with the topical facial cream applied as per the study protocol. Measurements adhere to a structured schedule to characterize the cream's impact on skin density.

SECONDARY OUTCOMES:
Assessment of Stinging Response to Topical Facial Cream Using Lactic Acid Stinging Test | Single assessment at Baseline (Day 0)
  This study evaluates cutaneous stinging response through a standardized Lactic Acid Stinging Test. Participants receive 10% lactic acid versus distilled water (control) applications on bilateral nasolabial folds. Stinging intensity is scored as: 0 (None), 1 (Mild), 2 (Moderate), 3 (Severe). Primary outcome: total score summation from both application sites.
Participant Self-Assessment of Facial Skin Condition Following Topical Product Application | Self-assessment questionnaires administered at Baseline (Day 0), Day 7, and Day 28 during 28-day intervention
  Participants assess facial skin condition using a validated self-assessment questionnaire. Assessment area: Full face. Scoring scale: 0 (ideal skin) to 9 (very unsatisfactory condition).
Participant-Reported Satisfaction with Topical Facial Product Efficacy. | Self-assessment questionnaires administered at Day 7 and Day 28 post-intervention initiation.
  Participants report satisfaction and perceived efficacy using a self-assessment questionnaire applied to full facial skin. Scale anchors: 1 (very dissatisfied) to 7 (very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- SGS-CSTC Standards Technical Services (Qingdao) Co., Ltd., Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No